CLINICAL TRIAL: NCT01263938
Title: Pilot Study to Evaluate Effects of Atorvastatin on Monocyte Activation in HAART-treated HIV Infected Individuals
Brief Title: Modulation of Monocyte Activation by Atorvastatin in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB Protocol #: 812196; P30AI045008 (NIH)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: HIV Dementia
Keywords: HIV; monocytes; CD16+; statins; mcp1; inflammation
MeSH Terms: conditions — AIDS Dementia Complex; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atorvastatin (Other)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — For subjects on PI-based HAART therapy: 10mg/day X 2weeks followed by 20mg/day.
  For subjects on non PI-based HAART therapy: 20mg/day X 2weeks followed by 40mg/day.
  Other Names: Lipitor

SUMMARY:
Activated monocytes play a key role in the pathogenesis of HIV-associated neurocognitive disorders (HAND). Individuals with HAND have expanded populations of activated monocytes. These monocytes are thought to emigrate into the CNS, where they produce neurotoxic proinflammatory factors, and also carry virus into the CNS. Statins are cholesterol lowering drugs with pleiotropic immunomodulatory / anti-inflammatory properties that are currently being explored for immunomodulation of T cell activation in several diseases, in addition to their established role to treat hyperlipidemia and atherosclerosis. The investigators in vitro data suggests that these drugs can downregulate monocyte activation patterns seen in HIV infection. No in vivo studies have yet been carried out to assess the effects of statins on the pro-inflammatory monocyte population in chronic HIV disease. This will be a pilot study of whether statin treatment will reduce the inflammatory monocyte phenotype and downregulate the inflammatory cytokines that have been linked to neuropathogenesis in HIV infection. If so, they may have potential as adjunctive therapy in HIV-associated neurological disease. The investigators propose to:

* Determine the effect of Atorvastatin on peripheral blood monocyte populations in a 12-week pilot study in chronically HIV-infected people on HAART therapy.
* Determine the relationship between changes in monocyte phenotype following Atorvastatin treatment, and soluble markers of activation/inflammation linked to neuropathogenesis, as well as activation status of T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HIV-1 infected individuals presently on HAART with no change in drug combination for at least 3 months at time of enrollment
2. Plasma viral load <200 copies / ml for at least 6 months prior to enrollment in the study
3. CD4 T cell count more than 350/ul
4. Willingness to use a method of contraception during the study period
5. Willingness to have blood drawn
6. If female, willingness to undergo pregnancy testing on a monthly basis and are not breastfeeding
7. Ability to understand and willingness to sign the informed consent
8. hs-CRP levels above the upper limit of normal (>3mg/L)

Exclusion Criteria:

1. Concomitant use of fibric acid derivatives or other lipid lowering agents including patients on statins and Ezetimibe
2. Use of any anti-inflammatory drugs (OTC or prescription) on a daily basis
3. Pregnancy or breast feeding
4. Active drug use or alcohol abuse/dependence, which in the opinion of the investigators will interfere with the patient's ability to participate in the study
5. Allergy or hypersensitivity to statins or any of its components
6. History of myositis or rhabdomyolysis with use of any statins
7. Patients who are on concurrent immunomodulatory agents, including systemic corticosteroids will be ineligible for 3 months after completion of therapy with the immunomodulating agents
8. History of inflammatory muscle disease such as poly or dermatomyositis
9. Serious intercurrent illness requiring systemic treatment and/or hospitalization within 30 days of entry
10. Evidence of active opportunistic infections requiring treatment or neoplasms that require chemotherapy during the study period
11. Creatine phosphokinase elevations (CPK) greater than 3 times the upper limit of normal
12. Known active liver disease or AST/ALT greater than 2x the upper limit of normal
13. Renal insufficiency, indicated by serum creatinine 2 mg/dl
14. Absolute neutrophil count (ANC) 1000/mm3, hemoglobin < 10.0 g/dL for males and <9 g/dL for females, platelet count 100,000/mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Collman, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the AIDS Clinical Trial Unit (ACTU) at the Hospital of University Of Pennsylvania, Philadelphia, PA. The screening and recruitment process was carried out during the period September 2011 thru April 2012.
Pre-assignment Details: Enrolled participants were assigned to treatment groups based on the nature of HAART therapy (PI- or non-PI based).
Period: Overall Study
Arm/Group | Atorvastatin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was an open label treatment study where enrolled participants at T=12wks post-drug treatment were compared to themselves at T=0 (pre-drug treatment), to assess changes in outcome measures as a result of treatment.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 3
  Race: Caucasian | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Monocyte Surface Markers Expression (Expressed as Percentage), Following Treatment of Chronic HIV+/ HAART+ Subjects With Atorvastatin (T=12wks Versus T=0wk).
Description: Effects of Atorvastatin on immune activation associated surface markers (CD16, CD163 and CCR2) of monocytes were assessed in chronic HIV+/HAART+ subjects following 12 weeks of treatment. Whole blood drawn from these subjects were stained with fluorochrome tagged antibodies to the surface markers. Stained whole blood cells were then acquired on a flow cytometer and analyzed using the Flowjo software to determine the percentage of cells (monocytes) expressing the specific marker. This was done before starting and after completing drug treatment to assess the effect of drug.
Time Frame: Subjects enrolled in the study following the screening visit were assessed for the primary outcome measures at T=0 (drug intervention begins); T=12wks (intervention ends)
Population: 1) Percentage of peripheral blood monocyte surface markers: CD16, CD163, CCR2
Measure: Mean (Standard Deviation); unit: Change T=0 to T=12 (percentage change)
Groups:
- Atorvastatin: For subjects on PI-based HAART:
  10mg/day X 2weeks followed by 20mg/day.
  For subjects on non PI-based HAART:
  20mg/day X 2weeks followed by 40mg/day.
  For all subjects treatment was stopped at 12 weeks.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 5
Change T=0 to T=12 (percentage change)
  Total CD14+CD16+ monocytes | 1.5 (10.2)
  CD14+CD163+ monocytes | -4.4 (18)
  CD14+CCR2+ monocytes | 0.5 (7.5)
Statistical Analysis 1: Comparison: Atorvastatin; Sample size calculations were based on having sufficient power to detect a change in each of the outcome variables from baseline to week 12.The effect size was calculated as (detectable difference in change in outcome) / (SD of the change). Based on preliminary in vitro data, the smallest effect size was 1.88. Assuming that only 40% of this effect will be present in vivo (effect size=0.75), alpha = 0.05 and 80% power, n=16 is needed to complete the study; Test type: Other; p = 0.625, Wilcoxon signed rank — Threshold for statistical significance: p<0.05
Statistical Analysis 2: Comparison: Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.813, Wilcoxon signed rank — Threshold for statistical significance: p<0.05
Statistical Analysis 3: Comparison: Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.999, Wilcoxon signed rank — Threshold for statistical significance: p<0.05

2. Primary Outcome: Change From Baseline in Levels of Plasma Inflammatory Marker MCP-1 of Chronic HIV+/ HAART+ Subjects.
Description: Monocyte specific inflammatory soluble factor MCP-1 was measured by ELISA in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following atorvastatin treatment.
Time Frame: as for outcome 1
Population: Plasma MCP-1 levels
Measure: Mean (Standard Deviation); unit: pg/ml (Change from T0 to T12)
Groups:
- Atorvastatin: For subjects on PI-based HAART:
  10mg/day X 2weeks followed by 20mg/day.
  For subjects on non PI-based HAART:
  20mg/day X 2weeks followed by 40mg/day.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 5
pg/ml (Change from T0 to T12) | 10 (176.5)
Statistical Analysis 1: Comparison: Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.999, Wilcoxon signed rank — Threshold for statistical significance: p<0.05

3. Primary Outcome: Change From Baseline in Levels of Plasma Inflammatory Marker sCD14 of Chronic HIV+/ HAART+ Subjects.
Description: Monocyte specific inflammatory soluble factor sCD14 was measured by ELISA in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following atorvastatin treatment.
Time Frame: as for outcome 1
Population: Plasma sCD14 levels
Measure: Mean (Standard Deviation); unit: ug/ml (Change fromT=0 to T=12wk)
Arm/Group | Atorvastatin
Number analyzed (Participants) | 5
ug/ml (Change fromT=0 to T=12wk) | -0.22 (0.7)
Statistical Analysis 1: Comparison: Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.813, Wilcoxon signed rank — Threshold for statistical significance: p<0.05

4. Primary Outcome: Change From Baseline in Levels of Plasma Inflammatory Marker sCD163 of Chronic HIV+/ HAART+ Subjects.
Description: Monocyte specific inflammatory soluble factor sCD163 was measured by ELISA in plasma of HIV+/HAART+ subjects at baseline and at 12 weeks following atorvastatin treatment.
Time Frame: as for outcome 1
Population: Plasma sCD163 levels
Measure: Mean (Standard Deviation); unit: ng/ml (Change fromT=0 to T=12wk)
Arm/Group | Atorvastatin
Number analyzed (Participants) | 5
ng/ml (Change fromT=0 to T=12wk) | -18 (81)
Statistical Analysis 1: Comparison: Atorvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.625, Wilcoxon signed rank — Threshold for statistical significance: p<0.05

ADVERSE EVENTS:
Time Frame: Data was collected over a period of sixteen weeks.
Description: To determine whether an adverse event had occurred or not, regular laboratory testing as well as investigator assessment was carried out during the Study period.
Arm/Group | Atorvastatin
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This study had a very small sample size of 5 subjects. Therefore due to lack of power the data is inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT01263938/Prot_SAP_000.pdf